CLINICAL TRIAL: NCT04639466
Title: Phase 1/2 Dose Escalation Study To Evaluate the Safety and Biologically Effective Dose of GEO-CM04S1, a Synthetic MVA-based SARS-CoV-2 Vaccine, Administered as One or Two Injections or as a Booster to Healthy Adult Volunteers
Brief Title: A Synthetic MVA-based SARS-CoV-2 Vaccine, GEO-CM04S1, for the Prevention of COVID-19 Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GeoVax, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20447; NCI-2020-08335 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20447 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-11-04; First posted 2020-11-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: COVID-19 Infection
MeSH Terms: conditions — COVID-19 | interventions — COH04S1 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Phase I Arm I (COH04S1) (Experimental): Participants receive COH04S1 IM in the non-dominant upper arm on day 0 and day 28 in the absence of unacceptable toxicity.
  Interventions: Biological: Synthetic MVA-based SARS-CoV-2 Vaccine COH04S1
- Phase I Arm II (COH04S1, placebo) (Active Comparator): Participants receive COH04S1 IM in the non-dominant upper arm on day 0 and placebo IM in the non-dominant upper arm on day 28 in the absence of unacceptable toxicity.
  Interventions: Drug: Placebo Administration; Biological: Synthetic MVA-based SARS-CoV-2 Vaccine COH04S1
- Phase I Arm III (placebo) (Placebo Comparator): Participants receive placebo IM in the non-dominant upper arm on day 0 and day 28 in the absence of unacceptable toxicity.
  Interventions: Drug: Placebo Administration
- Phase II Arm I (low dose COH04S1 booster) (Experimental): Participants receive low dose COH04S1 booster IM in non-dominant upper arm on day 1 in the absence of unacceptable toxicity.
  Interventions: Biological: Synthetic MVA-based SARS-CoV-2 Vaccine COH04S1
- Phase II Arm II (high dose COH04S1 booster) (Experimental): Participants receive high dose COH04S1 booster IM in non-dominant upper arm on day 1 in the absence of unacceptable toxicity.
  Interventions: Biological: Synthetic MVA-based SARS-CoV-2 Vaccine COH04S1

INTERVENTIONS:
Drug: Placebo Administration — Given IM in the non-dominant upper arm
  Arms: Phase I Arm II (COH04S1, placebo); Phase I Arm III (placebo)
Biological: Synthetic MVA-based SARS-CoV-2 Vaccine COH04S1 — Given IM in the non-dominant upper arm
  Other Names: COH04S1; SARS-CoV-2 Vaccine COH04S1; sMVA-based SARS-CoV-2 Vaccine COH04S1; GEO-CM04S1
  Arms: Phase I Arm I (COH04S1); Phase I Arm II (COH04S1, placebo); Phase II Arm I (low dose COH04S1 booster); Phase II Arm II (high dose COH04S1 booster)

SUMMARY:
This phase I trial evaluates the side effects and best dose of GEO-CM04S1 (previously designated as COH04S1), a synthetic modified vaccinia Ankara (MVA)-based SARS-CoV-2 vaccine, for the prevention of COVID-19 infection. COVID-19 infection is caused by the SARS-CoV-2 virus. SARS-CoV-2 has demonstrated the capability to spread rapidly, leading to significant impacts on healthcare systems and causing societal disruption. GEO-CM04S1 was created by placing small pieces of SARS-CoV-2 DNA (the chemical form of genes) into synthetic MVA, which may be able to induce immunity (the ability to recognize and fight against an infection) to SARS-CoV-2. The purpose of the Phase 1 study is to determine the safety and the optimal dose of the GEO-CM04S1 vaccine.

The Phase 2 study is designed as a multi-center, double-blind, randomized, parallel, study to evaluate the safety profile of 2 dose levels of GEO-CM04S1 as a single booster shot to assess the immune response measured by the fold-increase in antibody against SARS-CoV-2 Spike protein at day 28 post-injection among healthy adult volunteers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Safety and tolerability of the synthetic MVA-based SARS-CoV-2 vaccine GEO-CM04S1 vaccine at three different dose levels (DL): 1.0x10^7 plaque-forming unit (PFU)/dose, 1.0x10^8 PFU/dose, and 2.5x10^8 PFU/dose. (Phase I)

II. Evaluate the safety profile of a single-dose vaccine boost at day 7 post-injection of GEO-CM04S1. (Phase II)

III. Determine whether the GEO-CM04S1 dose levels tested (1.0x10^7 or 1.0x10^8) generate promising immune responses (>5-fold increase of Spike IgG over baseline) after single-dose booster injection, and select a promising dose to use for further study. (Phase II)

SECONDARY OBJECTIVES:

I. Longitudinal evaluation of humoral immunity. (Phase I)

II. Quality and properties of cellular and humoral immunity elicited as a result of the vaccination. (Phase I)

III. Explore the role of two injections versus one injection, and evaluate a placebo group. (Phase I)

III. Evaluate T cell-based antigen-specific immune responses at day 28 post-injection of single-dose GEO-CM04S1 vaccine boost. (Phase II)

IV. Evaluate SARS-CoV-2 S and N-specific Th1 vs Th2 polarization. (Phase II)

V. Assess levels of SARS-CoV-2 neutralizing antibodies and their activity against variants of concern (VOC) or variants of high consequence (VHC). (Phase II)

VI. Estimate the durability of antibody-based immune responses in a 12-month time period. (Phase II)

VII. Estimate the durability of T-cell-based immune responses in a 12-month time period. (Phase II)

VIII. Estimate the incidence of COVID-19 Moderate and Severe disease during follow-up (12 months). (Phase II)

IX. Evaluate the potential relationship between duration of immunity and COVID infection (incidence) over the 12-month study period. (Phase II)

X. Summarize outcomes, primary and secondary endpoints, based on pre-study mRNA vaccine received. (Phase II)

EXPLORATORY OBJECTIVES:

I. Surveillance for incidental coronavirus disease 2019 (COVID-19) infection during follow-up (1 year). (Phase I)

II. Quality and properties of cellular and humoral immunity elicited as a result of the vaccination. (Phase I)

III. Evaluate activated/cycling, cytotoxic/helper, and memory phenotype markers. (Phase II)

IV. Estimate SARS-CoV-2-specfic serum IgA and IgG over time. (Phase II)

OUTLINE: This is a dose-escalation study.

PHASE I: Participants are randomized to 1 of 3 arms.

ARM I: Participants receive GEO-CM04S1 intramuscularly (IM) in the non-dominant upper arm on day 0 and day 28 in the absence of unacceptable toxicity.

ARM II: Participants receive GEO-CM04S1 IM in the non-dominant upper arm on day 0 and placebo IM in the non-dominant upper arm on day 28 in the absence of unacceptable toxicity.

ARM III: Participants receive placebo IM in the non-dominant upper arm on day 0 and day 28 in the absence of unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 arms.

ARM I: Participants receive low dose GEO-CM04S1 booster IM in non-dominant upper arm on day 1 in the absence of unacceptable toxicity.

ARM II: Participants receive high dose GEO-CM04S1 booster IM in non-dominant upper arm on day 1 in the absence of unacceptable toxicity.

During Phase 1, participants are followed up at 7, 14, 28, 35, 42, 56, 90, 120, 180, 270, and 365 days. During Phase 2, participants are followed up at 7, 14, 28, 80, and 365 days.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I: Documented informed consent of the participant
* PHASE I: Age: >= 18 years and < 55 years
* PHASE I: Ability to read and understand English, Spanish, or Mandarin for consenting
* PHASE I: Platelets >= 100,000/mm^3 (within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE I: White blood cells (WBCs) 3,600-10,100/mm^3 (within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE I: Total bilirubin < 1.1 x upper limit of normal (ULN) (within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE I: Aspartate aminotransferase (AST) < 1.5 x ULN (within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE I: Alanine aminotransferase (ALT) < 1.5 x ULN (within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE I: Alkaline phosphatase (AP) < 1.1 x ULN (within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE I: Blood urea nitrogen (BUN) < 1.25 x ULN (within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE I: Creatinine less than or equal to the ULN (within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE I: Sodium 137-145 mEq/L (within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE I: Potassium 3.5-5.1 mEq/L (within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE I: Carbon dioxide 22-30 mmol/L (within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE I: Glucose 80-128 mg/dL (within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE I: Albumin 3.5-5.0 g/dL (within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE I: Hemoglobin (HGB) > 10.5 gm/dL (within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE I: Hematocrit (Hct) (within 30 days prior to day 0 of protocol therapy unless otherwise stated)

  * For females: 34.5-44.6 %
  * For males: 37.6-47.2 %
* PHASE I: Seronegative for human immunodeficiency virus (HIV) antigen (Ag)/antibody (Ab) combo, hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative) (within 30 days prior to day 0 of protocol therapy unless otherwise stated)

  * If positive, hepatitis C ribonucleic acid (RNA) quantitation must be performed
* PHASE I: History negative for COVID-19 and nasopharyngeal test results pending for SARS-CoV2 performed at City of Hope (COH) on nasal wash samples using the Diasorin Simplexa test (within 30 days prior to day 0 of protocol therapy unless otherwise stated)

  * Baseline SARS-CoV2serologic test will be performed at TGen using the InBios assay; the result will not be required for eligibility
* PHASE I: A documented electrocardiogram (ECG) and cardiac troponin must be within normal institutional limits in the past 30 days; "normal ECG with sinus tachycardia" or "normal ECG with sinus bradycardia" is allowable based on a history of absent cardiac/exercise related symptoms as determined by the principal investigator (P.I.) in consultation with a senior staff cardiologist (within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE I: Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (within 30 days prior to day 0 of protocol therapy unless otherwise stated)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* PHASE I: Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 weeks after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* PHASE II: Prior COVID-19 mRNA vaccination with EUA or FDA-approved vaccine, >= 6 months prior
* PHASE II: ECOG performance score 0-1
* PHASE II: Documented informed consent of the participant
* PHASE II: Age: >= 18 years
* PHASE II: Platelets >= 100,000/mm^3 (performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE II: WBCs 3,600-10,100/mm^3 (performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE II: Total bilirubin < 1.1 X ULN (performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE II: AST < 1.5 x ULN (performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE II: ALT < 1.5 x ULN (performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE II: AP < 1.1 x ULN (performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE II: BUN < 1.25 x ULN (performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE II: Creatinine less than or equal to the ULN (performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE II: Sodium 137-145 mEq/L (performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE II: Potassium 3.5-5.1 mEq/L (performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE II: Carbon dioxide 22-30 mmol/L (performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE II: Glucose 80-128 mg/dL (performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE II: Albumin 3.5-5.0 g/dL (performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE II: HGB > 10.5 gm/dL (performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* PHASE II: Hematocrit (Hct) (performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)

  * For females: 34.5-44.6 %
  * For males: 37.6-47.2 %
* PHASE II: Seronegative for HIV Ag/Ab combo, HCV, active HBV (Surface Antigen Negative) (performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)

  * If positive, hepatitis C RNA quantitation must be performed
* PHASE II: Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)

  * If the urine pregnancy test is inconclusive a serum pregnancy test will be required
* PHASE II: Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 weeks after the booster

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* PHASE I: Participants at increased risk of exposure to SARS-CoV-2, such as patient-facing health care workers and emergency responders are excluded
* PHASE I: Participants who would be at higher risk for severe COVID-19 according to known risk factors are excluded e.g. type 2 diabetes, obesity (body mass index [BMI] >= 35), congestive heart failure (New York Heart Association class >= I), history of coronary artery disease, or chronic obstructive pulmonary disease
* PHASE I: Participants using investigational or licensed agents that may prevent or treat SARS-CoV-2 are excluded
* PHASE I: Participants are excluded, who have any history of allergic diatheses as defined by a history of asthma, anaphylaxis, or generalized urticaria, or by daily use of antihistamines, episodic (more than once in past 3 months) inhalational medications including steroidal agents, non-steroidal agents, or cromolyn sodium
* PHASE I: Any previous condition, or one that becomes known during the screening period, which would suggest that the technicians and health professionals involved in the study would be exposed to specific infectious risk
* PHASE I: Surgery in past 6 months that required general anesthesia. Minor procedures, such as dental surgery and superficial diagnostic biopsies, are permitted
* PHASE I: Taking daily medications for chronic or intercurrent illness. Medications excluded from this rule are: thyroid replacement, estrogen replacement, dietary vitamins and protein supplements, mild anti-depressant and anxiety medication, and any medication not known or likely to be immunosuppressive, as determined by the P.I.
* PHASE I: Participants who have had a live vaccine =< 30 days prior to administration of study vaccine or subjects who are =< 2 weeks within administration of inactivated vaccines (e.g. influenza vaccine). Flu shots are allowed > 2 weeks before the first injection and > 2 weeks post 2nd injection
* PHASE I: Treatment with medication for high cholesterol or other lipid abnormality. Prophylactic medication is acceptable
* PHASE I: History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* PHASE I: History of adverse event with a prior smallpox vaccination
* PHASE I: Any previous condition, or one that becomes known during the screening period, that would suggest that the individual could be immunologically impaired, or for which this study would pose a danger to him/herself or about which the P.I., in evaluating the subject for eligibility, determines that this exclusion is appropriate
* PHASE I: Participants are excluded who have history of cancer other than basal cell skin cancer, or any condition, psychiatric or otherwise, that would preclude informed consent, consistent follow-up or compliance with any aspect of the study (e.g., untreated schizophrenia or other significant cognitive impairment, etc. as determined by the P.I.)
* PHASE I: Participants with severe migraine headaches (more than one per month on average in the past 6 months or requiring preventive medication) are excluded but those on effective medication (less than one migraine per month) are allowed to enroll
* PHASE I: History of heart disease, e.g. previous treated arrhythmia or myocardial infarction
* PHASE I: Horizontal positioning- induced or activities of normal living exercise-induced shortness of breath
* PHASE I: History of stroke or claudication
* PHASE I: Any of the following cardiac findings of ECG abnormality: 1) conduction disturbance (complete left or right bundle branch block, intraventricular conduction disturbance with QRS > 120 ms, atrioventricular block [AV] block of any degree, and corrected QT [QTc] prolongation > 450 msec for men and > 460 msec for women); 2) repolarization (ST segment or T wave) abnormality; 3) significant atrial or ventricular arrhythmia, including frequent ectopy (e.g., 2 premature ventricular contractions in a row); and 4) evidence of past myocardial infarction.
* PHASE I: Poxvirus vaccine in the last 12 months
* PHASE I: Any MVA vaccine or poxvirus vaccine in the last 12 months
* PHASE I: Any previous SARS-CoV-2 vaccine
* PHASE I: History of or prior treatment for diabetes type 1 or diabetes type 2; BMI < 18 or > 35. BMI can be rounded to the nearest integer
* PHASE I: Clinically significant uncontrolled illness
* PHASE I: Active infection requiring treatment
* PHASE I: Known history of immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection
* PHASE I: Diagnosis which has been associated with immunodeficiency
* PHASE I: Females only: Pregnant or breastfeeding
* PHASE I: Men with partners of child-bearing potential and women of children-bearing potential who are not willing to use medically effective birth control methods, e.g. contraceptive pill, condom, or diaphragm, and continue this for 6 weeks after the second and last dose of vaccine
* PHASE I: Participants who are employed by or are a student at City of Hope and are in a chain of command that reports directly to persons listed on the protocol as principal investigator or co-investigators; or are relatives or partners of the investigators
* PHASE I: Any other condition that would, in the investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns with clinical study procedures
* PHASE I: Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)
* PHASE I: Anyone considered to be in a vulnerable population as defined in 45 CFR 46.111 (a)(3) and 45 CFR 46, Subparts B-D
* PHASE II: Participants who would be at higher risk for severe COVID-19 according to known risk factors are excluded e.g. type 2 diabetes, obesity (BMI > 35), congestive heart failure (New York Heart Association Class >= I), history of coronary artery disease, cardiomyopathies, sickle cell disease, smoking, chronic kidney disease, immunocompromised state from solid organ transplant, or chronic obstructive pulmonary disease, or active cancers other than basal cell skin cancer at discretion of the investigator.
* PHASE II: Participants are excluded, who have any history of allergic diatheses as defined by a history of asthma, anaphylaxis, or generalized urticaria, episodic (more than once in past 3 months) inhalational medications including steroidal agents, non-steroidal agents, or cromolyn sodium
* PHASE II: Any previous condition, or one that becomes known during the screening period, which would suggest that the technicians and health professionals involved in the study would be exposed to specific infectious risk
* PHASE II: Taking daily medications for chronic or intercurrent illness. Medications excluded from this rule are: thyroid replacement, estrogen replacement, dietary vitamins and protein supplements, mild anti-depressant and anxiety medication, and any medication not known or likely to be immunosuppressive, as determined by the P.I.
* PHASE II: Participants who have had a live vaccine =< 30 days prior to administration of study vaccine or participants who are =< 2 weeks within administration of inactivated vaccines (e.g. influenza vaccine). Flu shots are allowed > 2 weeks before the booster injection and > 2 weeks post booster injection
* PHASE II: Intensive cytotoxic therapies, B- or T-cell depleting therapies, or checkpoint inhibitors within 30 days of enrollment
* PHASE II: Systemic corticosteroids required for chronic conditions at doses > 0.5 mg/kg/day prednisone equivalent within 14 days of enrollment
* PHASE II: Previously received a COVID-19 vaccine booster injection
* PHASE II: History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* PHASE II: History (suspected or confirmed) of myocarditis or pericarditis
* PHASE II: History of adverse event with a prior smallpox vaccination
* PHASE II: Any previous condition, or one that becomes known during the screening period, that would suggest that the individual could be immunologically impaired, or for which this study would pose a danger to him/herself or about which the P.I., in evaluating the participant for eligibility, determines that this exclusion is appropriate.
* PHASE II: Participants are excluded who have any condition, psychiatric or otherwise, that would preclude informed consent, consistent follow-up or compliance with any aspect of the study (e.g., untreated schizophrenia or other significant cognitive impairment, etc. as determined by the P.I.)
* PHASE II: Participants with severe migraine headaches (more than one per month on average in the past 6 months or requiring preventive medication) are excluded but those on effective medication (less than one migraine per month) are allowed to enroll.
* PHASE II: History of heart disease, e.g. previous treated arrhythmia or myocardial infarction
* PHASE II: History of stroke or claudication.
* PHASE II: Any MVA vaccine or poxvirus vaccine in the last 12 months;
* PHASE II: Clinically significant uncontrolled illness
* PHASE II: Active infection requiring treatment
* PHASE II: Females only: Pregnant or breastfeeding
* PHASE II: Men with partners of child-bearing potential and women of children-bearing potential who are not willing to use medically effective birth control methods, e.g. contraceptive pill, condom, or diaphragm, and continue this for 60 days after the second and last dose of vaccine;
* PHASE II: Persons listed on the protocol as Principal Investigator or Co-Investigators, and those who have disclosed a Conflict of Interest regarding COH04S1. Prospective participants who are COH employees reporting to study personnel conducting consent for the Phase 2 study must be consented by other consenting personnel to ensure no coercion. COH employees who would be involved in a quality or risk management function (auditing or monitoring) or the Study Management Team (SMT) with respect to this trial are ineligible.
* PHASE II: Any other condition that would, in the Investigator's judgment, contraindicate the participant's participation in the clinical study due to safety concerns with clinical study procedures.

Noncompliance

* PHASE II: Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).
* PHASE II: Anyone considered to be in a vulnerable population as defined in 45 CFR §46.111 (a)(3) and 45 CFR §46, Subparts B-D

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (Phase I) | Up to 365 days
  Evaluated based on the Division of Microbiology and Infectious Diseases criteria.
Incidence of adverse events (Phase II) | Within the first 7 days following booster injection
  Evaluated based on the Division of Microbiology and Infectious Diseases criteria.
Antibody levels to SARS CoV-2 Spike protein (Phase II) | Up to 365 days
  Assessed by Ortho VITROS Anti-SARS-CoV-2 IgG Quantitative assay.
Fold increase of Spike IgG levels (Phase II) | At 28 days post-injection

SECONDARY OUTCOMES:
Humoral immunity (Phase I) | During 1 year of observation
  Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)-specific IgA, IgG, and IgM measured in serum and saliva by enzyme-linked immunosorbent assay.
Level of SARS-CoV-2-specfic neutralizing antibodies (Phase I) | Up to 365 days
  Measure the generation of neutralizing antibodies in participants, and test whether they prevent infection of a susceptible cell line with a pseudo-type of the SARS-CoV-2 virus.
Th1 vs Th2 polarization (Phase I) | Up to 365 days
  SARS-CoV-2-specific IFN-gamma, TNF-alpha, IL-2, IL-4, IL6, IL-13 cytokine levels will be measured to assess Th1 vs Th2 polarization.
SARS-CoV-2- antigen specific T cell responses to the COH04S1 vaccine (Phase I) | Up to 365 days
  Assessed using overlapping peptide libraries specific for SARS-CoV-2.
Evolution of activated/cycling and memory phenotype markers on the surface of SARS-CoV-2- specific T cells elicited as a result of the COH04S1 vaccination (Phase I) | Up to 365 days
Comparison of immunogenicity and adverse events (Phase I) | Up to 365 days
  Immunogenicity and adverse events will be compared between one injection versus two injection groups.
T lymphocyte production of cytokines in response to in vitro stimulation with overlapping peptide libraries specific for SARS-CoV-2 (Phase II) | Up to 365 days
SARS-CoV-2-S and -N specific IFNγ (Th1) and IL-4 (Th2) cytokine levels (Phase II) | Up to 365 days
Neutralizing Ab levels (Phase II) | Up to 365 days
  Assessed by ability to prevent infection of a susceptible cell line with Spike pseudo-typed lentivirus representing different SARS-CoV-2 variants.
Antibody to SARS CoV-2 Spike protein (Phase II) | Up to 365 days
  Assessed by ORTHO VITROS assay, as well as antibody to N protein, and S protein neutralizing antibodies.
T lymphocyte production of cytokines in response to in vitro peptide library stimulation (Phase II) | Up to 365 days
COVID-19 disease that is moderate, severe, or critical (Phase II) | Up to 365 days
  Confirmed by polymerase chain reaction (PCR) viral load by Food and Drug Administration (FDA) guidelines February (Feb) 2021.
Confirmed COVID-19 infection by PCR viral load (Phase II) | Up to 365 days
Moderna or Pfizer vaccine received previously (Phase II) | Up to 365 days

OTHER OUTCOMES:
Incidence of coronavirus 2019 (COVID-19) infection (Phase I) | Up to 365 days
  Any incidental COVID-19 infection will be recorded occurring during the study follow-up period. The SARS-CoV-2-specific immune correlates of infected subjects will be compared with those uninfected.
Severity of COVID-19 and resolution (Phase I) | Up to 365 days
  Will be summarized descriptively to address concerns related to the potential for vaccine-induced disease enhancement.
Incidence of COVID-19 in placebo group (Phase I) | Up to 365 days
  Will be summarized to provide initial data on acquired COVID-19 infections in the same time period and subject pool.
SARS-CoV-2-specific neutralizing antibodies (Phase I) | Up to 365 days
In depth analysis of Th1 (IFN-gamma, TNF-alpha, IL-2)/Th2 (IL-4, IL-6, IL-13) cytokine expression via intracellular cytokine staining on selected samples (Phase I) | Up to 365 days
Phenotype markers on the surface of antigen specific T cells elicited as a result of the COH04S1 vaccination (Phase II) | Up to 365 days
  Will evaluate activated/cycling, cytotoxic/helper, and memory phenotype markers.
SARS-CoV-2-specfic IgA and IgG (Phase II) | Up to 365 days
  Measured in serum by enzyme-linked immunosorbent assay (ELISA) during 12 months of observation.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Principal Investigator — GeoVax, Inc.
Locations (3):
- United States (3):
  - EmVenio Research, Claremont, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Millennium Clinical Trials, Thousand Oaks, California